CLINICAL TRIAL: NCT07035249
Title: A Prospective, Single-Arm Clinical Trial Evaluating DCSZ11 Combined With Standard-of-Care Therapy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: DCSZ11 in Combination With Standard Therapy in Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD，professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025（648）
Record Dates: First submitted 2025-06-15; First posted 2025-06-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: DCSZ11; Solid Tumors; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: This single-center, open-label, single-arm trial employs a dose-escalation framework to assess DCSZ11's safety and biological activity when co-administered with guideline-directed standard therapy in advanced solid tumor patients. All participants will maintain fixed chemotherapy/immunotherapy regimens specific to their malignancy, with sole dose variation occurring for DCSZ11.
  Three subjects in the lead-in cohort will initiate DCSZ11 at 600 mg triweekly. Sequential cohorts will escalate to 800 mg and 1200 mg administered Q3W. The 800 mg tier derives from prior clinical evidence (NCT05785754) evaluating DCSZ11-pembrolizumab combinations. Incorporation of the 600 mg cohort facilitates refined escalation protocols and enhanced resolution in safety/tolerability profiling.
  Dose-limiting toxicities (DLTs) will undergo surveillance through a 21-day monitoring window. Escalation decisions will implement the Bayesian Optimal Interval (BOIN) methodology, with DLT classifications adhering to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): DCSZ11 at Low Dose in combination with the available standard treatment.
  Interventions: Drug: Low Dose DCSZ11; Drug: Standard Treatment
- Medium Dose (Experimental): DCSZ11 at Medium Dose in combination with the available standard treatment.
  Interventions: Drug: Medium Dose DCSZ11; Drug: Standard Treatment
- High Dose (Experimental): DCSZ11 at High Dose in combination with the available standard treatment.
  Interventions: Drug: High Dose DCSZ11; Drug: Standard Treatment

INTERVENTIONS:
Drug: Low Dose DCSZ11 — Patients will receive DCSZ11 at 600 mg every three weeks (Q3W).
  Arms: Low Dose
Drug: Medium Dose DCSZ11 — Patients will receive DCSZ11 at 800 mg Q3W.
  Arms: Medium Dose
Drug: High Dose DCSZ11 — Patients will receive DCSZ11 at 1200 mg Q3W.
  Arms: High Dose
Drug: Standard Treatment — The available standard treatment for head and neck cancer patients.

SUMMARY:
To evaluate the safety and efficacy of DCSZ11 in combination with standard therapy in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years.
2. Willing and able to provide written informed consent for the study.
3. Patients with histologically confirmed advanced or metastatic solid tumors. Note: Patients must have guideline-eligible standard chemotherapy and immunotherapy options available.Patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) must have PD-L1 Combined Positive Score (CPS) ≥1.Lung cancer patients with known actionable driver gene mutations/genomic aberrations (e.g., EGFR sensitizing mutations, BRAF V600E mutation, ROS1 rearrangements, NTRK gene fusions, ALK rearrangements) are excluded.Prior adjuvant or neoadjuvant chemotherapy is permitted, provided ≥6 months have elapsed between the last dose of chemotherapy/immunotherapy and documented recurrent disease.Gastric cancer patients must be HER2-negative.
4. Patients must have at least one measurable lesion per RECIST 1.1 criteria. Lesions located in previously irradiated areas may be considered measurable if there is objective evidence of progression in those lesions prior to study enrollment.
5. Patients with previously treated central nervous system (CNS) metastases are eligible provided they meet all the following criteria:

   1. Stability (i.e., no evidence of progression on magnetic resonance imaging [MRI]) for ≥4 weeks prior to the first dose of study drug, and
   2. All neurological symptoms have returned to baseline, and
   3. No requirement for steroid therapy for at least 14 days prior to the first dose of study intervention.

   Patients with signs or symptoms suggestive of CNS metastases must undergo brain imaging within 2 weeks prior to the first dose of study drug to confirm the absence of detectable CNS disease.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate organ function and bone marrow reserve per laboratory assessments within 10 days prior to first study drug administration:

   1. Bone marrow function:

      * Absolute neutrophil count (ANC) ≥1,500/µL
      * Hemoglobin ≥9 g/dL (must be achieved without erythropoietin dependency AND without packed red blood cell [pRBC] transfusion within the preceding 2 weeks)
      * Platelet count ≥100,000/µL
   2. Hepatic function:

      * Total serum bilirubin ≤1.5 × upper limit of normal (ULN); or direct bilirubin ≤ULN for patients with total bilirubin >1.5 × ULN
      * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN if liver metastases present)
   3. Renal function:

      * Estimated creatinine clearance ≥30 mL/min (per Cockcroft-Gault formula)
8. PD-L1 status must be available for all patients via approved immunohistochemistry assay.
9. Resolution of all prior treatment-related toxicities to Grade ≤1 or baseline, or determination as irreversible sequelae.

   *Note: Grade ≤2 neuropathy and/or hearing loss, alopecia of any grade, or autoimmune endocrinopathies on stable replacement therapy are permitted.*
10. Female patients must agree to refrain from breastfeeding for 5 months after last study dose and satisfy one of:

    1. Postmenopausal for ≥1 year prior to screening, or
    2. Surgically sterile, or
    3. Agreement to use one highly effective contraceptive method plus one additional barrier method from signing informed consent form (ICF) until 5 months after last study dose, or
    4. Practice true abstinence* when consistent with preferred lifestyle Periodic abstinence, withdrawal, spermicide-only, or lactational amenorrhea are unacceptable. Female/male condoms must not be used concomitantly.
11. Male patients, even surgically sterilized (i.e., post-vasectomy), must agree to either:

    1. Use effective barrier contraception from ICF signing until 2 months after last DCSZ11 dose, or
    2. Practice true abstinence* when consistent with preferred lifestyle Exclusions as per Criterion 10.
12. Willingness and ability to comply with scheduled visits and procedures per protocol.

Exclusion Criteria:

1. Systemic anticancer therapy or investigational products within 6 months prior to first study dose.

   *Note: Low-dose corticosteroids (oral prednisolone ≤10 mg daily or equivalent) and therapy with bisphosphonates or RANK ligand (RANKL) inhibitors are permitted.*
2. Extensive radiotherapy (RT) ≤6 months prior to treatment initiation (*≤7 days for palliative local RT outside chest/brain*) OR unresolved RT-related toxicity requiring corticosteroids.
3. Second primary malignancy within 3 years, except:

   Adequately treated basal cell/locally confined squamous skin cancer Localized prostate cancer Carcinoma in situ of cervix/breast Resected colorectal adenomatous polyps Other malignancies not requiring active anticancer therapy.
4. Known active CNS metastases and/or carcinomatous meningitis.
5. Major surgery within 4 weeks or minor surgery within 2 weeks prior to first dose.

   All wounds must be fully healed without infection/dehiscence, with full recovery and no ongoing surgical complications.
6. Known hypersensitivity to any component of the study drug(s).
7. Prior immunotherapy discontinued due to:

   Grade ≥3 immune-related adverse events (irAEs) (except endocrinopathies controlled with replacement) Grade 2 myocarditis OR recurrent Grade 2 pneumonitis.
8. Active autoimmune disease requiring systemic immunosuppression within 2 years. Exempt: Physiologic hormone replacement (thyroxine, insulin, corticosteroids for adrenal/pituitary insufficiency).
9. Immunodeficiency diagnosis OR chronic systemic steroids (>10 mg prednisolone-equivalent/day) or other immunosuppressants within 7 days prior to first dose.
10. History of lung RT >30 Gy within 6 months prior to treatment.
11. History of (non-infectious) pneumonitis/interstitial lung disease (ILD) requiring steroids OR current pneumonitis/ILD.
12. History of allogeneic tissue/solid organ transplantation.
13. Live/live-attenuated vaccines within 4 weeks prior to treatment initiation. Inactivated vaccines permitted.
14. Active infection requiring systemic therapy.
15. Hepatitis B surface antigen (HBsAg)-positive with detectable HBV DNA.
16. Hepatitis C virus (HCV) infection with detectable HCV RNA at screening.
17. History within ≤6 months prior to first dose of:

    NYHA Class III/IV congestive heart failure

    Unstable angina

    Myocardial infarction

    Symptomatic ischemic heart disease

    Uncontrolled hypertension despite optimal therapy

    Persistent symptomatic arrhythmia >Grade 2

    Pericardial effusion/restrictive cardiomyopathy. Permitted: Chronic atrial fibrillation on stable anticoagulation.
18. Any condition compromising informed consent, confounding results, or limiting protocol compliance-including medical/psychiatric/social factors-that, per investigator judgment, contraindicates participation.
19. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The ratio of participants assessed with complete response (CR) or partial response(PR) as a best overall response.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 years
  The ratio of subjects assessed with CR or PR or stable disease (SD) as a best overalresponse.
DRR (Durable Response Rate) | 2 years
  DRR is defined as the proportion of objective response (CR and PR as determined by the investigator) lasting at least 6 months at any time within 12 months of initiation of treatment.
DOR (Duration of Response) | 2 years
  DOR is defined as the time from the date when the PR is first recorded or better to the date when the disease progression is first recorded (for the responder, i.e., PR or better). Responders who did not record disease progress will be censored on the date that the last assessment was SD or better.
TTR (Response Time） | 2 years
  TTR is defined as the time from the date of the first administration to the date of the first record of the objective tumor response (CR and PR determined by the investigator).
PFS (progression-free survival) | 2 years
  PFS is defined as the duration until disease progression or death in participants fromthe first dose of immunization.
OS (Overall Survival) | 2 years
  0S is defined as the duration until death in participants from the first dose ofimmunization.
TTP (Time to Progression) | 2 years
  TTP is defined as the time from the date of first dose to the date of first documented disease progression, as defined by standard disease criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Professor, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilgus TA, Bergdall VK, Tober KL, Hill KJ, Mitra S, Flavahan NA, Oberyszyn TM. The impact of cyclooxygenase-2 mediated inflammation on scarless fetal wound healing. Am J Pathol. 2004 Sep;165(3):753-61. doi: 10.1016/S0002-9440(10)63338-X. PMID 15331400
- [Background] Barbera S, Nardi F, Elia I, Realini G, Lugano R, Santucci A, Tosi GM, Dimberg A, Galvagni F, Orlandini M. The small GTPase Rab5c is a key regulator of trafficking of the CD93/Multimerin-2/beta1 integrin complex in endothelial cell adhesion and migration. Cell Commun Signal. 2019 May 28;17(1):55. doi: 10.1186/s12964-019-0375-x. PMID 31138217
- [Background] Blackburn JWD, Lau DHC, Liu EY, Ellins J, Vrieze AM, Pawlak EN, Dikeakos JD, Heit B. Soluble CD93 is an apoptotic cell opsonin recognized by alphax beta2. Eur J Immunol. 2019 Apr;49(4):600-610. doi: 10.1002/eji.201847801. Epub 2019 Feb 7. PMID 30656676
- [Background] Sun Y, Chen W, Torphy RJ, Yao S, Zhu G, Lin R, Lugano R, Miller EN, Fujiwara Y, Bian L, Zheng L, Anand S, Gao F, Zhang W, Ferrara SE, Goodspeed AE, Dimberg A, Wang XJ, Edil BH, Barnett CC, Schulick RD, Chen L, Zhu Y. Blockade of the CD93 pathway normalizes tumor vasculature to facilitate drug delivery and immunotherapy. Sci Transl Med. 2021 Jul 28;13(604):eabc8922. doi: 10.1126/scitranslmed.abc8922. PMID 34321321
- [Background] Wu B, Fu L, Guo X, Hu H, Li Y, Shi Y, Zhang Y, Han S, Lv C, Tian Y. Multi-omics profiling and digital image analysis reveal the potential prognostic and immunotherapeutic properties of CD93 in stomach adenocarcinoma. Front Immunol. 2023 Jan 25;14:984816. doi: 10.3389/fimmu.2023.984816. eCollection 2023. PMID 36761750
- [Background] Lugano R, Vemuri K, Yu D, Bergqvist M, Smits A, Essand M, Johansson S, Dejana E, Dimberg A. CD93 promotes beta1 integrin activation and fibronectin fibrillogenesis during tumor angiogenesis. J Clin Invest. 2018 Aug 1;128(8):3280-3297. doi: 10.1172/JCI97459. Epub 2018 Jun 25. PMID 29763414
- [Background] Langenkamp E, Zhang L, Lugano R, Huang H, Elhassan TE, Georganaki M, Bazzar W, Loof J, Trendelenburg G, Essand M, Ponten F, Smits A, Dimberg A. Elevated expression of the C-type lectin CD93 in the glioblastoma vasculature regulates cytoskeletal rearrangements that enhance vessel function and reduce host survival. Cancer Res. 2015 Nov 1;75(21):4504-16. doi: 10.1158/0008-5472.CAN-14-3636. Epub 2015 Sep 11. PMID 26363010
- [Background] Dieterich LC, Mellberg S, Langenkamp E, Zhang L, Zieba A, Salomaki H, Teichert M, Huang H, Edqvist PH, Kraus T, Augustin HG, Olofsson T, Larsson E, Soderberg O, Molema G, Ponten F, Georgii-Hemming P, Alafuzoff I, Dimberg A. Transcriptional profiling of human glioblastoma vessels indicates a key role of VEGF-A and TGFbeta2 in vascular abnormalization. J Pathol. 2012 Nov;228(3):378-90. doi: 10.1002/path.4072. Epub 2012 Aug 31. PMID 22786655
- [Background] Khan KA, Naylor AJ, Khan A, Noy PJ, Mambretti M, Lodhia P, Athwal J, Korzystka A, Buckley CD, Willcox BE, Mohammed F, Bicknell R. Multimerin-2 is a ligand for group 14 family C-type lectins CLEC14A, CD93 and CD248 spanning the endothelial pericyte interface. Oncogene. 2017 Nov 2;36(44):6097-6108. doi: 10.1038/onc.2017.214. Epub 2017 Jul 3. PMID 28671670
- [Background] Jain RK. Antiangiogenesis strategies revisited: from starving tumors to alleviating hypoxia. Cancer Cell. 2014 Nov 10;26(5):605-22. doi: 10.1016/j.ccell.2014.10.006. Epub 2014 Nov 10. PMID 25517747
- [Background] Reichart PA, Philipsen HP. Oral erythroplakia--a review. Oral Oncol. 2005 Jul;41(6):551-61. doi: 10.1016/j.oraloncology.2004.12.003. Epub 2005 Apr 9. PMID 15975518
- [Background] Boucher Y, Kumar AS, Posada JM, Gjini E, Pfaff K, Lipschitz M, Lako A, Duda DG, Rodig SJ, Hodi FS, Jain RK. Bevacizumab improves tumor infiltration of mature dendritic cells and effector T-cells in triple-negative breast cancer patients. NPJ Precis Oncol. 2021 Jun 29;5(1):62. doi: 10.1038/s41698-021-00197-w. PMID 34188163